CLINICAL TRIAL: NCT05451329
Title: A Phase 2, Double-masked, Randomized, Vehicle-controlled, Dose-response Study Assessing the Safety and Ocular Hypotensive Efficacy of VVN539 in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension
Brief Title: A Phase 2 Double-masked Study of VVN539 in Subjects With Elevated Intraocular Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VivaVision Biotech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVN539-CS-201
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Double-masked, randomized, parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VVN539 Ophthalmic Solution 0.02% (Active Comparator): VVN539 Ophthalmic Solution 0.02%
  Interventions: Drug: VVN539 Ophthalmic Solution 0.02%
- VVN539 Ophthalmic Solution 0.04% (Active Comparator): VVN539 Ophthalmic Solution 0.04%
  Interventions: Drug: VVN539 Ophthalmic Solution 0.04%
- VVN539 Ophthalmic Solution Vehicle (Placebo Comparator): VVN539 Ophthalmic Solution Vehicle
  Interventions: Drug: VVN539 Ophthalmic Solution Vehicle

INTERVENTIONS:
Drug: VVN539 Ophthalmic Solution 0.02% — Once a day [q.d.] in the morning, q.d. in the evening and twice a day [b.i.d.]) will be tested for 7-9 days
  Arms: VVN539 Ophthalmic Solution 0.02%
Drug: VVN539 Ophthalmic Solution 0.04% — Once a day [q.d.] in the morning, q.d. in the evening and twice a day [b.i.d.]) will be tested for 7-9 days
  Arms: VVN539 Ophthalmic Solution 0.04%
Drug: VVN539 Ophthalmic Solution Vehicle — Once a day [q.d.] in the morning, q.d. in the evening and twice a day [b.i.d.]) will be tested for 7-9 days
  Arms: VVN539 Ophthalmic Solution Vehicle

SUMMARY:
This is a prospective, parallel-comparison, multi-center, double-masked, randomized, vehicle-controlled dose-response study assessing the safety and ocular hypotensive efficacy of VVN539 in subjects with POAG or OHT. Three different dosing regimens (once a day [q.d.] in the morning, q.d. in the evening and twice a day [b.i.d.]) will be tested for 7-9 days, each.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Diagnosis of primary open-angle glaucoma or ocular hypertension in both eyes that are untreated, or if treated, in the opinion of the investigator are well controlled on 2 or fewer ocular hypotensive medications prior to Visit 1.
* Unmedicated intraocular pressure of ≥ 22 mm Hg and ≤ 36 mm Hg in the study eye, with no more than 5 mm Hg inter-eye difference at 08:00AM and 10:00AM at Visit 2.
* Corrected visual acuity in each eye +1.0 or better by Early Treatment Diabetic Retinopathy Scale in each eye (equivalent to Snellen 20/200)

Exclusion Criteria:

* Known hypersensitivity to any kinase inhibitors, any excipient or preservative of the formulation or to topical anesthetics or fluorescein.
* Unmedicated IOP of > 36 mm Hg in either eye at any time point at Visit 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Yan Li, M.D., Study Director — VivaVision
Locations (1):
- Lexitas, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VVN539 Ophthalmic Solution 0.02% | VVN539 Ophthalmic Solution 0.04% | VVN539 Ophthalmic Solution Vehicle
Started | 23 | 22 | 23
Completed | 20 | 20 | 23
Not Completed | 3 | 2 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Investigational Product Lot exchange | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VVN539 Ophthalmic Solution 0.02% | VVN539 Ophthalmic Solution 0.04% | VVN539 Ophthalmic Solution Vehicle | Total
Number analyzed (Participants) | 23 | 22 | 23 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 9 | 23
  >=65 years | 18 | 13 | 14 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (9.0) | 65.1 (13.4) | 64.7 (16.4) | 66.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 12 | 33
  Male | 11 | 13 | 11 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 3 | 11
  Not Hispanic or Latino | 17 | 20 | 20 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 18 | 19 | 23 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 23 | 68

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure
Description: mmHg
Time Frame: 8AM, 10AM, and 4PM at Day 7; Day 14 and Day 21
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | VVN539 Ophthalmic Solution 0.02% | VVN539 Ophthalmic Solution 0.04% | VVN539 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 23 | 22 | 23
mmHg
  0800 AM Day 7 | 21.8 (4.6) | 20.5 (2.5) | 23.4 (3.9)
  1000 AM Day 7 | 19.7 (4.7) | 19.0 (2.8) | 22.0 (3.1)
  0400 PM Day 7 | 19.1 (4.1) | 18.1 (2.6) | 21.7 (2.9)
  0800 AM Day 14 | 21.1 (5.0) | 19.6 (3.9) | 23.1 (3.5)
  1000 AM Day 14 | 19.9 (5.1) | 18.2 (4.3) | 22.1 (3.0)
  0400 PM Day 14 | 19.7 (5.2) | 18.0 (2.8) | 22.0 (3.9)
  0800 AM Day 21 | 19.7 (3.6) | 19.2 (2.8) | 23.4 (3.9)
  1000 AM Day 21 | 19.2 (5.0) | 19.1 (3.3) | 22.6 (3.2)
  0400 PM Day 21 | 18.7 (5.2) | 18.8 (3.0) | 21.7 (3.7)

2. Secondary Outcome: Mean Change in Intraocular Pressure From Baseline
Description: mmHg
Time Frame: 8AM, 10AM, and 4PM at Day 7; Day 14 and Day 21
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | VVN539 Ophthalmic Solution 0.02% | VVN539 Ophthalmic Solution 0.04% | VVN539 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 23 | 22 | 23
mmHg
  0800 AM Day 7 | -3.6 (4.1) | -4.1 (2.7) | -2.0 (2.8)
  1000 AM Day 7 | -5.3 (4.2) | -5.0 (3.0) | -2.3 (3.0)
  0400 PM Day 7 | -3.3 (3.5) | -4.6 (2.6) | -1.3 (2.2)
  0800 AM Day 14 | -4.3 (4.3) | -5.0 (4.0) | -2.2 (2.7)
  1000 PM Day 14 | -5.1 (4.2) | -5.8 (3.6) | -2.1 (2.3)
  0400 PM Day 14 | -2.7 (4.6) | -4.8 (3.3) | -0.9 (3.5)
  0800 AM Day 21 | -5.7 (2.7) | -5.4 (2.8) | -2.0 (3.3)
  1000 AM Day 21 | -5.7 (3.9) | -5.0 (3.7) | -1.5 (2.4)
  0400 PM Day 21 | -3.7 (4.3) | -3.9 (2.8) | -1.2 (3.4)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | VVN539 Ophthalmic Solution 0.02% | VVN539 Ophthalmic Solution 0.04% | VVN539 Ophthalmic Solution Vehicle
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 11/23 | 10/22 | 1/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VVN539 Ophthalmic Solution 0.02% (N=23) | VVN539 Ophthalmic Solution 0.04% (N=22) | VVN539 Ophthalmic Solution Vehicle (N=23)
Conjunctival hyperaemia (Eye disorders) | 11 (11) | 10 (10) | 1 (1)
Ocular hyperaemia (Eye disorders) | 3 (3) | 5 (5) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 3 (3) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All investigators will work collaboratively with the Sponsor on presentations and publications.

DOCUMENTS (2):
  • Study Protocol (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT05451329/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT05451329/SAP_001.pdf